CLINICAL TRIAL: NCT04711330
Title: Response and Toxicity Prediction by Microbiome Analysis After (Concurrent) Chemo RT in Locally Advanced NSCLC Treated With IO (Durvalumab)
Brief Title: Response and Toxicity Prediction by Microbiome Analysis After (Concurrent) Chemoradiotherapy
Acronym: Prediction
Status: Active, not recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: The Netherlands Cancer Institute (Other); Jessa Hospital (Other)
Responsible Party: Principal Investigator, pbaas, Professor, Leiden University Medical Center
Other Study IDs: 76017
Record Dates: First submitted 2021-01-12; First posted 2021-01-15 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-03

CONDITIONS: Non Small Cell Lung Cancer Stage III; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Collection of bacterial specimen from throat and feces.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with maintenance immunotherapy after concurrent chemo/RT: Observation of response and response. The microbiome of the patients throat and stool will be analyzed before the standard treatment with IO is initiated after completion of the chemoradiation therapy.
  No intervention is planned.

SUMMARY:
The predictive value of the microbiome (throat swabs, stool and of bronchial samples) to identify patients who will relapse during durvalumab treatment after CRT (False negative Rate) at 6 months. Exploratory endpoints include the effects of antibiotic therapy before and during IO treatment on toxicity and response rate. The role of exhaled breath analysis in prediction of response and toxicity will also be investigated.

DETAILED DESCRIPTION:
In this observational study we aim to investigate the predictive value of the microbiome (throat swabs and stool) to identify patients who will relapse during durvalumab treatment after CRT (False negative Rate) at 6 months.

Collection of stool and throat swipe before start of durvalumab treatment; sampling of blood and exhaled air for analysis of volatile organic compounds.

Improved clinical outcomes after adjuvant treatment with durvalumab following concurrent chemoradiotherapy (CCRT) for locally advanced NSCLC (PACIFIC trial), led to the rapid adoption of this treatment strategy as standard of care. However, despite the improved progression free survival and overall survival, recurrence rate remains high. Approximately 45% of patients will relapse within 1 year, despite adjuvant durvalumab therapy. To date no performant biomarker predicting treatment response or failure nor toxicity exists and the number of prospective studies addressing this issue is limited. Both PD-L1 TPS and TMB should be considered 'enriching' parameters improving response-chances, but they are far from an ideal biomarker. Non-invasive biomarkers are essential in the future for better patient selection and therapy allocation. One of the potential non-invasive biomarkers of interest is the microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Stages IIIA, IIIB and IIIC (as per UICC 8th TNM edition) NSCLC (histologically or cytologically confirmed) amenable for durvalumab treatment after sequential or concurrent chemoradiotherapy according to local standards. Patients that received neoadjuvant/adjuvant chemotherapy for surgically treated stages I to III NSCLC are allowed as long as therapy was completed at least 6 months prior to the diagnosis of disease recurrence amenable for chemoradiotherapy and resolution of all treatment related toxicity ≤ grade 1 .
2. No signs of disease progression after CCRT
3. At least 1 cycle of chemotherapy before or concurrent during radiotherapy but no more chemotherapy between last radiotherapy session and start durvalumab
4. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
5. Absence of any of following targetable driver mutations: EGFR, ALK, ROS1
6. over 18 years
7. ECOG 0-1
8. Must be willing to provide collected stool samples and allow to obtain a throat swab during the observation period. A pulmonary protected brush swab will only be optionally performed in a selected number of patients.
9. Demonstrate adequate organ function

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Has had prior monoclonal antibody therapy within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
3. Previous treatment with PD-1-PD-L1 axis inhibiting immunotherapy.
4. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, anti-phospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis with the following exceptions:

   * Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.
   * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
   * Skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic immunosuppressive treatment, in particular corticosteroids are permitted to enrol.
5. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids, and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
6. Subjects who have undergone organ transplant or allogeneic stem cell transplantation.
7. Active malignancy or a prior malignancy within the past 3 years, with the following exceptions:

   * Patients with completely resected basal cell carcinoma, cutaneous squamous cell carcinoma, cervical carcinoma in-situ, breast carcinoma in-situ, and patients with isolated elevation in prostate-specific antigen or low risk prostate cancer (managed with watchful waiting) are allowed.
   * Patients who underwent mediastinal radiotherapy in the past are not allowed.
8. Subjects with chronic infections/infectious disorders (eg. Clostridium colitis)
9. Have known but untreated driver mutations of the EGFR gene or ALK or ROS1 translocation.
10. Has evidence of symptomatic interstitial lung disease or an active, non-infectious pneumonitis.
11. Has an active chronic infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who will receive durvalumab as standard of care after completion of (concurrent) chemo-radiation therapy for stage III non small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-02 (Estimated)

PRIMARY OUTCOMES:
Prediction of outcome (progression) based on microbiome analysis | 1 year
  To investigate the predictive value of the microbiome (throat swabs and stool) to identify patients who will relapse during durvalumab treatment after CRT (False negative Rate) at 6 months

SECONDARY OUTCOMES:
Prediction of toxicity based on microbiome analysis | 1 year
  To investigate the predictive value of the microbiome (throat swabs and stool ) to identify patients that develop irAE's during durvalumab treatment after CRT.
Prediction of outcome (disease controle rate) based on microbiome analysis | 1 year
  To determine disease control rate (DCR ie. Stable disease, partial response, and complete response) and PFS at 6 months and correlate to the microbiome.
Relationship between circulating immune cells and microbiome outcome | 1 year
  To investigate to what extend cytological characteristics of circulating immune cells obtained from responders and non-responders differ and to explore to what extend these differences relate to the microbiome.
Value of analysis of exhaled breath at 6 months | 6 months
  To investigate the predictive value of exhaled breath analysis (by eNose) to identify patients who will relapse or progress during durvalumab treatment after CRT (False negative Rate) at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Baas, MD PhD, Principal Investigator — Leiden University Medical Center
Locations (6):
- Belgium (4):
  - Kristof Cuppens, Hasselt, Flanders
  - Piet Verkouteren, Aalst
  - Ingel Demedts, Roeselare
  - Lynn Decoster, Turnhout
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam
  - Leiden University Medical center, Leiden

IPD SHARING:
Plan to Share IPD: Undecided
microbioma data from the participants

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT04711330/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT04711330/ICF_001.pdf